CLINICAL TRIAL: NCT03716687
Title: Prophylactic Negative Pressure Wound Therapy for High Risk Laparotomy Wounds. Randomized Prospective Clinical Trial.
Brief Title: Prophylactic Negative Pressure Wound Therapy for High Risk Laparotomy Wounds. A Randomized Prospective Clinical Trial.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No chance to enroll sufficient cases. Several coinvestigator centers have never started recruiting.
Sponsor: St. Borbala Hospital (Other Government)
Collaborators: Semmelweis University (Other); Department of Surgery, Jahn Ferend Dél-Pesti Kórház és Rendelőintézet, Budapest (Unknown); Department of Surgery, Somogy Megyei Kaposi Mór Oktatókórház, Kaposvár (Unknown); Institute of Surgery, University of Debrecen (Unknown); Department of Surgery, University of Szeged (Unknown); Department of Surgery, Uzsoki Utcai Kórház és Rendelőintézet, Budapest (Unknown); Department of Surgery, Markusovszky Egyetemi Oktatókórház, Szombathely (Unknown); Department of Surgery, Bács-Kiskun Megyei Kórház, Kecskemét (Unknown); Department of Surgery, Kenézy Gyula Egyetemi Oktatókórház, Debrecen (Unknown); Department of Surgery, Szent Rókus Kórház, Baja (Unknown); Department of Surgery, St. Borbala hospital, Tatabanya (Unknown)
Responsible Party: Principal Investigator, Dr. Balázs Bánky PhD, Head of the Department of Surgery, St. Borbala Hospital, St. Borbala Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OGYÉI/15347-9/2018
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Surgical Wound; Wound Dehiscence, Surgical; Surgical Site Infection; Dehiscence of Internal Surgical Wound
Keywords: negative pressure wound closure; surgical site infection; cost effectiveness
MeSH Terms: conditions — Surgical Wound; Surgical Wound Dehiscence; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: 50-50% randomisation into interventional (ciNPWT) and control (traditionaltreatment) groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ciNPWT (Experimental): Prophylactic negative pressure wound dress (Hartmann) is set up for 5 days right after operation.
  Continous -90 Hgmm negative pressure mode selected. No change of wound dress until 5 days completed.
  Interventions: Device: Prophylactic negative pressure wound dressing after laparotomy
- Traditional wound dressing (No Intervention): Control group with traditional, dry laparotomy wound dressing.

INTERVENTIONS:
Device: Prophylactic negative pressure wound dressing after laparotomy — Five days of -90 Hgmm continuous negative pressure wound dressing left on primary closed laparotomy wound.
  Arms: ciNPWT

SUMMARY:
Negative pressure wound closure technique (NPWT) has been widely introduced in different clinical settings. Most of the studies report it as an effective and cost-effective method to treat complicated surgical wounds or even open abdomen.

NPWT as a prophylactic effort to prevent complications of high risk surgical wounds has recently been introduced, but the concept is still lacking clinical evidence in terms of clinical effectiveness and cost effectiveness.

In this randomized, multi centric study investigators aim to compare prophylactic negative pressure wound closure (ciNPWT) with traditional, dry wound dressing at high infection risk laparotomy wounds.

DETAILED DESCRIPTION:
The aim is to compare ciNPWT (closed incisional negative pressure wound dress) technique to the traditional, dry wound dressing technique at high infection risk laparotomy wounds.

Control arm will be treated "as usual": sterile gauze or high-absorbing surgical wound dress.

Experimental arm will be dressed with: one layer of silver-containing, impregnated mesh laxer (Atrauman® Ag - Hartmann) directly placed on the primary closed wound, one layer of alcohol-soaked foam (VivanoMed® White Foam - Hartmann) and sufficient-size sealant film (Hydrofilm® - Hartmann).

A negative pressure of -90 Hgmm will be administered in a continuous mode over 5 days postoperatively.

Surgical site infection and abdominal wall dehiscence rate will be assessed, as well as cost effectiveness will be calculated at both arms.

ELIGIBILITY:
Inclusion Criteria:

* High risk laparotomy patients. SSI risk at least 3x higher than normal rate (6-8%)
* Surgical wound type III or IV..

Exclusion Criteria:

* Patients not giving informed consent.
* Patients requiring open abdominal wound care.
* Patients with abdominal wall malignancy,
* Patients with peritoneal carcinomatosis,
* Patients who are planned for second look laparotomy within 5 days,
* Patients with less thank 3 month life expectancy.
* Patients who are operated with existing wound infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection requiring wound re-opening (suture removal) and open wound treatment. (Clavien-Dindo 2)

SECONDARY OUTCOMES:
Full thickness abdominal wall dehiscence, requiring re-operation | 30 days
  Full thickness abdominal wall dehiscence, requiring re-operation

CONTACTS AND LOCATIONS:
Locations (1):
- St. Borbala Hospital, Tatabánya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sahebally SM, McKevitt K, Stephens I, Fitzpatrick F, Deasy J, Burke JP, McNamara D. Negative Pressure Wound Therapy for Closed Laparotomy Incisions in General and Colorectal Surgery: A Systematic Review and Meta-analysis. JAMA Surg. 2018 Nov 1;153(11):e183467. doi: 10.1001/jamasurg.2018.3467. Epub 2018 Nov 21. PMID 30267040
- [Result] Curran T, Alvarez D, Pastrana Del Valle J, Cataldo TE, Poylin V, Nagle D. Prophylactic closed-incision negative-pressure wound therapy is associated with decreased surgical site infection in high-risk colorectal surgery laparotomy wounds. Colorectal Dis. 2019 Jan;21(1):110-118. doi: 10.1111/codi.14350. Epub 2018 Aug 20. PMID 30047611
- [Result] Gachabayov M, You K, Sullivan R, Bergamaschi R. A Retrospective Cohort Study to Determine Predictive Factors for Abdominal Wound Disruption Following Colorectal Surgery. Ostomy Wound Manage. 2018 Apr;64(4):22-29. PMID 29718814
- [Result] Strugala V, Martin R. Meta-Analysis of Comparative Trials Evaluating a Prophylactic Single-Use Negative Pressure Wound Therapy System for the Prevention of Surgical Site Complications. Surg Infect (Larchmt). 2017 Oct;18(7):810-819. doi: 10.1089/sur.2017.156. Epub 2017 Sep 8. PMID 28885895
- [Result] Athanasiou AN, Spartalis M, Spartalis E. Prophylactic Negative Pressure Dressing Use in Closed Laparotomy Wounds After Abdominal Operations: What We Really Know? Ann Surg. 2018 Jul;268(1):e19-e20. doi: 10.1097/SLA.0000000000002413. No abstract available. PMID 28692475
- [Derived] Herczeg A, Szijarto A, Fulop A, Varga K, Marton J, Loderer Z, Mohos B, Pancel B, Szendrenyi V, Lazar G, Libor L, Kaposztas Z, Mathe E, Bursics A, Kecskedi B, Sikorszki L, Venczel L, Banky B. Prophylactic Negative Pressure Wound Therapy Reduces Superficial Surgical Site Infection Risk of Emergency Surgery Patients: Results of a Multicenter Randomised Prospective Clinical Trial. Int Wound J. 2025 Jul;22(7):e70718. doi: 10.1111/iwj.70718. PMID 40605477